## NAVAL MEDICAL RESEARCH COMMAND (NMRC) DEFENSE INFECTIOUS DISEASES DIRECTORATE (DIDD) TRANSLATIONAL AND CLINICAL RESEARCH (TraCR) DEPARTMENT

## Statistical Analysis Plan for PATH Protocol CVIA 088

#### **Study Title:**

Controlled Human Infection Model Challenge/Rechallenge: *Shigella flexneri* 2a and *S. sonnei* cross-protective antigens discovery in healthy adults in the United States

Version 1.0 04 October 2023

NCT Number: NCT04992520

### **CVIA 088 Statistical Analysis Plan Revision History**

| Version Number | Version Date | Summary of Changes |
|----------------|--------------|-----------------------|
| 1.0 | 04OCT2023 | N/A - initial version |

Version 1.0; 04OCT2023

2

#### **CVIA 088 Signature Page**

Protocol Number: CVIA 088 (version 4.2; dated 16 January 2023)

Statistical Analysis Plan (version 1.0)

#### **PATH Statistician**

Signed:

DocuSigned by:

Yuxiao Tang

Signer Name: Yuxiao Tang

Signing Reason: I approve this document Signing Time: 05-Oct-2023 | 07:08 PDT -01E3B2D8EC9547EA8EA3E82F09C8DA89

Yuxiao Tang, PhD

PATH, Center for Vaccine Innovation and Access (CVIA)

2201 Westlake Avenue, Suite 200

Seattle, WA 98121

#### Principal Biostatistician

DocuSigned by:

Chad Porter

Signed:

V

Signer Name: Chad Porter

Signing Reason: I approve this document Signing Time: 05-Oct-2023 | 07:16 PDT -1E303E02D6874702B5263ED08D55F532

1.0 01.0 1.077

Chad Porter, PhD, MPH

TraCR, NMRC

503 Robert Grant Avenue

Silver Spring, MD 20910

#### **Table of Contents**

| | | | _ |
|---|------|---------------------------------------------------------------|---|
| 1 | Abł | previations and Definitions | 6 |
| 2 | Pre | Pace | 7 |
| 3 | Intr | oduction | 7 |
| 4 | Stud | ly Objectives | 8 |
| | 4.1 | Primary Objective | 8 |
| | 4.2 | Secondary Objective | 8 |
| | 4.3 | Exploratory Objectives. | 8 |
| 5 | Stud | ly Endpoints | 8 |
| | 5.1 | Primary Endpoint | 8 |
| | 5.2 | Secondary Endpoints | 9 |
| 6 | Rea | ctogenicity Events | 9 |
| | 6.1 | Adverse Events (AEs) | 9 |
| | 6.2 | Suspected Adverse Reaction | 9 |
| | 6.3 | Solicited and Anticipated AEs | 0 |
| | 6.4 | AEs of Special Interest (AESI) | 0 |
| | 6.5 | Serious Adverse Events (SAEs) | 0 |
| | 6.6 | AE Relationship to the Investigational Product | 0 |
| | 6.7 | AE Safety Assessments | 0 |
| 7 | Stud | dy Methods1 | 0 |
| | 7.1 | Study Design and Plan | 0 |
| | 7.2 | Study Population | 0 |
| | 7.2. | 1 Selection of Participants | 0 |
| | 7.2. | 2 Inclusion and Exclusion Criteria1 | 0 |
| | 7.2. | Continuing Eligibility Criteria to Proceed to Cohort 1B or 2B | 0 |
| | 7.3 | Challenge Administration1 | 1 |
| | 7.3. | 1 Challenge Strains Administered | 1 |
| | 7.3. | 2 Method of Selecting Eligible Subjects for Second Challenge | 1 |
| | 7.3. | 3 Blinding1 | 1 |
| | 7.4 | Immunology Testing1 | 1 |
| 8 | San | nple Size Considerations | |

| 9 | Ge | neral | Study Considerations | 12 |
|---|---|---|---|---|
| ( | 9.1 | Safe | ety/Full Analysis Population | 12 |
| ( | 9.2 | Per- | -Protocol Population | 12 |
| ( | 9.3 | Imn | nunology Population | 13 |
| ( | 9.4 | Mis | ssing Data | 13 |
| ( | 9.5 | Out | come Adjudication | 13 |
| 10 | Pui | pose | of the Analyses | 13 |
| | 10.1 | Tim | ning of Analyses | 14 |
| | 10.2 | Safe | ety Evaluation | 14 |
| | 10. | 2.1 | Demographics and Other Baseline Characteristics | 14 |
| | 10. | 2.2 | Medical History | 14 |
| | 10. | 2.3 | Concomitant Medications | 15 |
| | 10. | 2.4 | Vital Signs and Physical Evaluations | 15 |
| | 10. | 2.5 | Safety Analyses | 15 |
| | 10.3 | Imn | nunogenicity Analyses | 15 |
| 11 | Ge | neral | Statistical Considerations | 17 |
| 12 | Rej | portir | ng Conventions | 17 |
| 13 | Tec | chnic | al Details | 17 |
| 14 | Ap | pendi | ices | 17 |
| | 14.1 | San | nple Data Tables and Figures for Final Clinical Study Report | 18 |
| | 14.2 | San | nple Data Tables and Figures for Exploratory Analyses | 33 |
| 15 | Ref | feren | ces | 75 |

#### 1 Abbreviations and Definitions

| AE | Adverse event |
|--------------|------------------------------------------------|
| AESI | |
| | Adverse event of special interest |
| ALS<br>ANOVA | Antibody in lymphocyte supernatant |
| | Analysis of variance |
| AR | Attack rate |
| ATC | Anatomical Therapeutic Chemical |
| cfu | Colony-forming units |
| cGMP | Current Good Manufacturing Practice |
| CHIM | Controlled human infection model |
| CI | Confidence interval |
| CRO | Contract research organization |
| CSR | Clinical study report |
| CVIA | Center for Vaccine Innovation and Access |
| DIDD | Defense Infectious Diseases Directorate |
| dL | Deciliter |
| ELISA | Enzyme-linked immunosorbent assay |
| GMFR | Geometric mean fold-rise |
| GMT | Geometric mean titer |
| Hg | Mercury |
| IBS | Irritable bowel syndrome |
| IgA | Immunoglobulin A |
| IgG | Immunoglobulin G |
| IQR | Interquartile range |
| LPS | Lipopolysaccharide |
| MedDRA® | Medical Dictionary for Regulatory Activities® |
| μg | Microgram |
| mg | Milligram |
| mL | Milliliter |
| NMRC | Naval Medical Research Command |
| PT | Preferred term |
| PSRT | Protocol Safety Review Team |
| PVT | Psychomotor vigilance test |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SBA | Serum bactericidal antibody |
| SOC | System organ class |
| SOP | Standard operating procedure |
| TD | Travelers' diarrhea |
| TLFs | Tables, listings, and figures |
| TraCR | Translational and Clinical Research Department |
| WHO | World Health Organization |
| WRAIR | Walter Reed Army Institute of Research |
| WINAIN | wanter Reed Army institute of Research |

#### 2 Preface

The purpose of this Statistical Analysis Plan (SAP) for the study entitled, "Controlled Human Infection Model Challenge/Rechallenge: *Shigella flexneri* 2a and *S. sonnei* cross-protective antigens discovery in healthy adults in the United States," (PATH protocol CVIA 088; ClinicalTrials.gov Identifier: NCT04992520) is to delineate a robust statistical analysis plan beyond the overview that is included in the study protocol (protocol v4.2; dated 16 January 2023).

This document describes all analyses planned for the study, as well as outlines sample tables, listings, and figures (TLFs) for the final analyses. Additionally, this document contains a review of the study design, general statistical considerations, and comprehensive statistical analysis methods for safety and immunogenicity outcomes. Deviations from this SAP will be described and justified in protocol amendments and/or in the clinical study report (CSR), as appropriate. The reader of this SAP is encouraged to review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

This SAP was completed following guidelines from the following PATH Standard Operating Procedure (SOP) documents:

- 1. SOP-00045: "Quality Control of Statistical Analysis" (version 1.0; dated 14 May 2021)
- 2. SOP-00046: "Development of Statistical Analysis Plans" (version 1.0; dated 14 May 2021)

#### 3 Introduction

Shigella is a leading cause of diarrhea-attributed morbidity and mortality globally. Shigella accounts for approximately 0.1 to 1.1 million deaths (60% in children under 5 years of age) and 90 to 165 million cases of dysentery annually [1-3]. Among travelers, Shigella are a cause of severe travelers' diarrhea (TD) [4]. In adults, shigellosis is linked to several post-infectious sequelae, including irritable bowel syndrome (IBS) and reactive arthritis [5-7]. Additionally, Shigella infection is associated with cognitive and physical stunting in children residing in low-income countries, which further highlights the pathogen's associated morbidity.

The *Shigella* controlled human infection model (CHIM) has been used to evaluate the efficacy of investigational *Shigella* vaccines since the studies of Shaughnessy and colleagues in 1946 among prison inmates in Joliet, Illinois [8]. Since then, CHIM trials evaluating *Shigella* vaccine candidates have been conducted at several sites in the United States, mostly with *S. flexneri* 2a (strain 2457T) [7, 9-11] and *S. sonnei* (strain 53G) [9, 10, 12], but also with wild-type and toxinminus mutants of *S. dysenteriae* type 1 [12-18].

This SAP is for a CHIM study designed to assess the cross-protection and markers of protection after challenge and rechallenge with heterologous serogroups of *Shigella*. In addition to assessing the potential reduction in shigellosis rates following heterologous rechallenge, efforts will be made to identify novel, cross-protective *Shigella* antigens that could enhance vaccine coverage among existing vaccines or serve as stand-alone subunit vaccines.

#### 4 Study Objectives

#### 4.1 Primary Objective

To evaluate the cross-species protection conferred by a rechallenge with a *Shigella* species of a different serotype.

#### 4.2 Secondary Objective

To determine effects of previous challenge when rechallenged with *Shigella* of a different serotype on stool output and clinical symptoms.

#### 4.3 Exploratory Objectives

- 1. To determine IgG and IgA responses to *Shigella* species-specific lipopolysaccharide (LPS) upon challenge or rechallenge.
- 2. To utilize novel analyses of immune responses, including antigen arrays, to identify protective immune responses in individuals protected from shigellosis upon challenge or rechallenge.
- 3. To identify potential protective antigens on the challenge organisms.
- 4. To confirm that the serum IgG to the O-antigen is a correlate of protection for shigellosis.
- 5. To assist in the development of international standards against *Shigella* antigens.
- 6. To measure mucosal and systemic immune responses to experimental infection.
- 7. To obtain and archive samples for future proteomics, inflammatory marker, microbiome, and/or transcriptomics and systems biology efforts based on the recently published consensus schedule and events table [19].
- 8. To evaluate the cognitive and sleep impact of acute diarrhea using psychomotor vigilance testing (PVT) and actigraphy.
- 9. To evaluate serum bactericidal antibody (SBA) titers against *S. flexneri* 2a 2457T and *S. sonnei* 53G (responders defined as ≥4-fold increase in SBA titer at designated time points post-initial challenge and heterologous rechallenge).
- 10. To evaluate the ability of wearable-collected data to predict clinical and/or microbiological endpoints.

#### 5 Study Endpoints

#### 5.1 Primary Endpoint

The primary endpoint for outcomes following initial challenge and heterologous rechallenge is the onset of shigellosis [20], defined as:

• Severe diarrhea: ≥6 loose (grade 3-5) stools within 24 hours or >800 grams of loose (grade 3-5) stools within any 24-hour window

OR

 Moderate diarrhea (4 to 5 loose stools within 24 hours or 401-800 grams of loose (grade 3-5) stools within 24 hours) with fever OR with one or more moderate constitutional or enteric symptom OR ≥2 episodes of vomiting within any 24-hour window

OR

• Dysentery: ≥2 loose stools with gross blood (hemoccult positive) in 24 hours AND fever OR ≥1 moderate constitutional/enteric symptom OR ≥2 episodes of vomiting in 24 hours

Fever: oral temperature ≥38°C confirmed within about 20 minutes

Constitutional/enteric symptoms: nausea, abdominal cramps/pain, myalgia, arthralgia, malaise

#### 5.2 Secondary Endpoints

Secondary endpoints for this study following initial challenge and heterologous rechallenge are:

- Maximum 24-hour stool output
- Percent of participants with severe diarrhea
- Percent of participants with diarrhea of any severity
- Total weight of grade 3-5 stools per participant
- Percent of participants with nausea, vomiting, anorexia, abdominal pain/cramps rated as moderate to severe
- Percent of participants who meet the definition of dysentery
- Mean/median time to onset of diarrhea
- Number of participants with more severe diarrhea (defined as  $\geq$ 10 loose [grade 3-5] stools within 24 hours or  $\geq$ 1000 grams of loose [grade 3-5] stools within 24 hours)
- Number of participants with fever
- Shigella clinical severity score post-challenge
- Number of colony-forming units (cfu) of the challenge strain per gram of stool

Note: Period of data collection for all secondary endpoints is during the inpatient period.

#### **6** Reactogenicity Events

#### 6.1 Adverse Events (AEs)

Information pertaining to AEs is detailed in Section XIII, part 5 of the study protocol.

#### **6.2** Suspected Adverse Reaction

Information pertaining to suspected adverse reactions is detailed in Section XIII, part 5 of the study protocol.

#### 6.3 Solicited and Anticipated AEs

Information pertaining to solicited and anticipated AEs is detailed in Section XIII, part 5 of the study protocol.

#### 6.4 AEs of Special Interest (AESI)

Information pertaining to AESIs is detailed in Section XIII, part 5 of the study protocol.

#### 6.5 Serious Adverse Events (SAEs)

Information pertaining to SAEs is detailed in Section XIII, part 5 of the study protocol.

#### 6.6 AE Relationship to the Investigational Product

Information pertaining to AE relationships to the investigational product is detailed in Section XIII, part 6 of the study protocol.

#### 6.7 AE Safety Assessments

Information pertaining to AE safety assessments is detailed in Section XIII, part 9 of the study protocol.

#### 7 Study Methods

#### 7.1 Study Design and Plan

Information pertaining to the study design and plan is detailed in Section VIII, parts 1 and 2 of the study protocol.

#### 7.2 Study Population

#### 7.2.1 Selection of Participants

Information pertaining to the selection of participants is detailed in Section IX, part 1 of the study protocol.

#### 7.2.2 Inclusion and Exclusion Criteria

Information pertaining to the inclusion and exclusion criteria is detailed in Section IX, parts 2 and 3 (respectively) of the study protocol.

#### 7.2.3 Continuing Eligibility Criteria to Proceed to Cohort 1B or 2B

Information pertaining to continuing eligibility criteria to proceed to cohort 1B or 2B is detailed in Section IX, part 4 of the study protocol.

#### 7.3 Challenge Administration

#### 7.3.1 Challenge Strains Administered

Participants will be challenged with approximately  $1.5 \times 10^3$  cfu of *S. flexneri* 2a strain 2457T or  $1.5 \times 10^3$  cfu of *S. sonnei* strain 53G.

S. flexneri 2a strain 2457T is a well-characterized Shigella strain that has had the greatest range of doses tested. This specific strain was isolated from a clinically ill patient in Japan in the early 1950s.

S. sonnei strain 53G has previously been used in low inoculum doses; however, a lyophilized preparation of this strain was recently manufactured to simplify the inoculum preparation process.

Both of these strains were manufactured under current Good Manufacturing Practice (cGMP) conditions at the Walter Reed Army Institute of Research (WRAIR) Pilot BioProduction Facility in Silver Spring, MD.

#### 7.3.2 Method of Selecting Eligible Subjects for Second Challenge

Information pertaining to the selection of eligible subjects for a second challenge is detailed in Section XV, part 2 of the study protocol.

#### 7.3.3 Blinding

As all subjects in each cohort will receive the same challenge strain, blinding will not be employed. However, the adjudication of clinical outcomes will be blinded to both strain and cohort. The study statistician and any other designated staff will have access to the unblinded cohort information and will assign new subject IDs that differs from those assigned at enrollment.

#### 7.4 Immunology Testing

During this study, samples will be collected from all subjects on pre-determined study days to complete the required immunological testing. The following tests will be completed during the study:

- 1. Serum IgG and IgA responses to *S. flexneri* 2a LPS, *S. flexneri* 2a Invaplex, IpaB, IpaC, and IpaD (2457T strain); *S. sonnei* LPS, *S. sonnei* Invaplex, IpaB, IpaC, and IpaD (53G strain)
- 2. Antibody in lymphocyte supernatant (ALS) responses to *S. flexneri* 2a LPS, *S. flexneri* 2a Invaplex, IpaB, IpaC, and IpaD (2457T strain); *S. sonnei* LPS, *S. sonnei* Invaplex, IpaB, IpaC, and IpaD (53G strain)
- 3. Fecal IgA responses to *S. flexneri* 2a LPS, *S. flexneri* 2a Invaplex, IpaB, IpaC, and IpaD (2457T strain); *S. sonnei* LPS, *S. sonnei* Invaplex, IpaB, IpaC, and IpaD (53G strain)
- 4. Salivary IgA responses to *Shigella* antigens (LPS, IpaB, IpaC, IpaD)

11

#### **8** Sample Size Considerations

Presuming a shigellosis rate of 70% in naïve participants, a sample size of 16 participants will yield a 95% confidence interval (asymptotic estimates) of 48-92%, while a sample size of 8 participants will yield a 95% confidence interval (asymptotic estimates) of 38-100%. Presuming an ability to pool naïve participants (if the cohorts have a comparable attack rate), a sample size of 19 participants in the previously *S. sonnei* 53G-challenged arm and 16 participants in the *S. flexneri* 2457T-naïve arm provides a >80% power to detect a shigellosis risk difference of 46% presuming a  $\geq$ 70% attack rate in *Shigella*-naïve participants, while a sample size of 11 participants in the previously *S. flexneri* 2457T-challenged arm and 8 participants in the *S. sonnei* 53G-naïve arm provides a >80% power to detect a shigellosis risk difference of 60% presuming a  $\geq$ 70% attack rate in *Shigella*-naïve participants (based on a Pearson's chi-squared test for proportional differences and a two-sided *alpha*=0.05). A power curve, corresponding to a sample size of 19 participants in the previously *S. sonnei* 53G-challenged arm and 16 participants in the *S. flexneri* 2457T-naïve arm and an attack rate of 70% in *Shigella*-naïve participants is below:



#### 9 General Study Considerations

#### 9.1 Safety/Full Analysis Population

All subjects who have been screened, consented, and proceeded to receive the challenge strain will serve as the primary analysis population for the safety endpoints. Adverse events will be listed individually and summarized by the Medical Dictionary for Regulatory Activities® (MedDRA®) body system and preferred terms within a body system for each study group. Serious and/or unexpected AEs will also be discussed on a case-by-case basis.

#### 9.2 Per-Protocol Population

The per-protocol population will consist of all subjects in the safety/full analysis population who have no major protocol violations that are determined to potentially interfere with the clinical

assessment. This population will serve as the primary analysis population for the primary and secondary endpoints. Membership in this study population will be determined in a blinded fashion.

#### 9.3 Immunology Population

Analyses will include both qualitative (responder rates) and quantitative results. All challenged subjects with collected post-challenge specimens relevant to each immunologic measure will be included in analyses. This population will serve as the primary analysis population for the immunogenicity endpoints.

#### 9.4 Missing Data

Although data are not anticipated to be missing during the inpatient phase of the study, the potential for subjects to be unable to collect a loose stool during a diarrheal episode could lead to missing data within the stool log and affect the primary endpoint. In this scenario, stools will be designated a weight of 0; however, if the adjudication committee determines that a subject should be characterized as having shigellosis, they would be included in analyses pertaining to that endpoint. Any other missing data due to subject-specific deviations (e.g., failure to return for follow-up or sample collection outside of the timeframe indicated in the protocol) will be documented. These data will be assumed to be missing at random and will be excluded from analyses unless they are identified as an outlier. If a data point is identified as an outlier, sensitivity analyses will be performed to assess the impact of including or excluding the outlier. Significant differences between these sensitivity analyses will be reported.

#### 9.5 Outcome Adjudication

Prior to the closeout of the study, detailed data on stool output and other clinical outcomes will be entered into Advantage eClinical and monitored. To obtain an unbiased determination of the study outcomes, an independent outcome adjudication committee will blindly evaluate challenge outcome data after completion of all inpatient phases of the study. To ensure a blinded review, new subject IDs that differ from those assigned at enrollment will be utilized.

If there are any individuals selected to participate in the challenge phase of the study that do not receive the investigational product, they will be excluded from the information presented. Additional information pertaining to the outcome adjudication committee is detailed in Section XIII, part 11 of the study protocol.

#### 10 Purpose of the Analyses

Analyses will focus on descriptive methods to estimate rates, measures of central tendency (e.g., means, medians, etc.), and data distributions (standard deviations, confidence intervals (CIs), interquartile ranges (IQRs), etc.).

Rates of solicited and unsolicited AEs will be tabulated by level of severity. All rates will be determined with two-sided exact 95% CIs.

During each day of the inpatient period, subjects will be monitored for loose stools (not meeting the diarrhea definition), diarrhea, dysentery, hypovolemia, nausea, vomiting, abdominal cramps/pain, fever, headache, anorexia, arthralgia, bloating, chills, constipation, flatulence, myalgia, lightheadedness, malaise, tenesmus, urgency, abdominal tenderness, abdominal distention, or otherwise abnormal abdominal exam.

Planned statistical evaluations are based on the proportion of subjects meeting prospectively-defined clinical, microbiological, and immunological endpoints. The shigellosis attack rate (AR) will be calculated for all study groups, using the standard definition of: (# with endpoint/# receiving inoculum) x 100%, along with 95% CIs (both asymptotic estimates and exact) for each study group. ARs between *Shigella*-naïve participants and previously challenged participants will be compared using a Pearson's chi-squared or Fisher's exact test, as appropriate. Summary tables will also be created to detail quantitative and temporal features of the illness, such as diarrheal stool frequency and volume, maximum temperature observed, and time to illness and infection. Continuous variables will be analyzed using nonparametric statistics unless assumptions are fulfilled for parametric statistics.

All statistical tests will be interpreted in a two-tailed fashion using an *alpha*=0.05.

#### 10.1 Timing of Analyses

Safety data will be prepared periodically and reviewed by the Protocol Safety Review Team (PSRT) throughout the trial.

After the completion of all inpatient phases of the study for all cohorts, blinded clinical outcome data will be prepared and reviewed by the outcome adjudication committee.

The full set of samples for key immunogenicity variables will be completed at the Day 180 visit.

A final analysis of all data collected will be performed after all data queries have been resolved, membership in the per-protocol population has been determined in a blinded fashion, and the database has been locked.

#### **10.2** Safety Evaluation

#### 10.2.1 Demographics and Other Baseline Characteristics

A summary table of continuous and categorical measures will be presented by study group and overall. A demographics listing will also be prepared, including information on sex, race, ethnicity, and age (in years).

#### **10.2.2** Medical History

Summaries of subjects' pre-existing medical conditions will be prepared; individual subject listings will also be prepared.

#### **10.2.3 Concomitant Medications**

Any medications that were taken either prior to or during the study will be coded according to the Anatomical Therapeutic Chemical (ATC) classification system using the World Health Organization (WHO) Drug Dictionary. Summaries as well as individual subject listings will be prepared.

#### 10.2.4 Vital Signs and Physical Evaluations

Systolic and diastolic blood pressure (mmHg), oral temperature (°F), and heart rate (beats/minute) will be obtained multiple times daily throughout the inpatient period and at designated study visits per the study schedule.

A complete physical exam will be conducted during the screening visit and on Day -2 or -1 as part of the screening process. Focused physical exams (symptom focused) will be conducted prior to receipt of any challenge product, daily during the inpatient stay, and as needed during the outpatient visits. A table summarizing the occurrence of abnormal physical exam findings will be presented by body system and study group.

#### 10.2.5 Safety Analyses

Table listings for AEs outlined in Section 6 of this SAP will be created to show the AE(s) a subject experiences, the onset date, the end date, the severity, the relationship to the challenge strain and/or antibiotic administration, and the outcome of the listed AE.

Additionally, all safety data will be listed individually and summarized by body system and preferred term within a body system for each study group. Serious and/or unexpected AEs will also be described on a case-by-case basis. For the tabulation of AEs by body system, a subject will be counted only once in a given body system. For example, a subject reporting nausea and diarrhea will be reported as one subject, but the symptoms will be listed as two separate AEs within the class. Therefore, the total number of AEs reported within a body system may exceed the number of subjects within the body system reporting AEs.

The proportion of all subjects with each AE will be summarized with a point estimate for percent and exact 95% CIs. Summary tables describing the number and percentage of subjects who experience each AE will be created. In addition, tables will be prepared to list each AE, the number of subjects experiencing an event at least once, and the proportion of subjects with an AE(s). AEs will be divided into defined severity grades (mild, moderate, severe, or potentially life threatening). The tables will also differentiate the relationship of AEs to the investigational product.

#### 10.3 Immunogenicity Analyses

Immunogenicity analyses will include both qualitative (responder rates) and quantitative (using log<sub>10</sub>-transformed values) outcomes.

Graphical displays of immune responses will include the following:

- 1. Scatter plots of peak fold-rise in antibody titer by study group for each antigen (serology and fecal IgA)
- 2. Salivary IgA responses
- 3. Response kinetics (group geometric mean titer [GMT] at each study time point to assess multiple dose effect)

Descriptive statistics (including mean and standard deviation of log<sub>10</sub> titers, GMT and 95% CIs, median, and IQR) will be tabulated by cohort, challenge status (initial challenge and secondary challenge), and time point. Geometric mean fold-rises (GMFRs) from baseline will also be calculated and summarized.

Between-group comparisons will be examined with nonparametric tests (Kruskal-Wallis test for continuous data and Fisher's exact test for categorical data), unless assumptions are fulfilled for ANOVA or Pearson's chi-squared test. Nonparametric paired t-tests (Wilcoxon paired signed-rank test) will be used to compare individual post-challenge to baseline responses within each study group, unless assumptions are fulfilled for paired t-tests. Comparisons of ALS responses post-challenge will be performed using the Kruskal-Wallis test. All statistical tests will be interpreted in a two-tailed fashion using *alpha*=0.05.

#### Immunologic Responder Definitions

Serology: An immunologic responder is defined as any subject who demonstrates a  $\geq$ 4-fold rise in reciprocal serum enzyme-linked immunosorbent assay (ELISA) antibody titers from baseline. A 4-fold rise is calculated by dividing the post-challenge reciprocal endpoint titer by the baseline reciprocal endpoint titer. All statistical analyses will be performed on  $\log_{10}$ -transformed titer values. Titers will be displayed graphically as  $\log_{10}$  reciprocal endpoint titers or geometric mean titers.

Antibody in Lymphocyte Supernatant (ALS): An immunologic responder is any subject who demonstrates a  $\geq$ 4-fold rise in reciprocal titers from baseline. A 4-fold rise is calculated by dividing the post-challenge reciprocal endpoint titer by the baseline reciprocal endpoint titer. Once a subject is defined as an 'immunologic responder', that person is permanently categorized as a 'RESPONDER'. All statistical analyses will be performed on  $\log_{10}$ -transformed titer values. Titers will be displayed graphically as  $\log_{10}$  reciprocal endpoint titers or geometric mean titers.

Fecal IgA: Total IgA content in the fecal extract samples will be determined by a modified ELISA method using commercial purified total IgA standard. Specimens with an IgA concentration  $<10 \mu g/mL$  will be excluded from all assessments of responder rates. Specific antibody levels in the fecal extracts will be determined using similar ELISA methods to those described above. Fecal antibodies will be reported as adjusted endpoint titers and calculated by dividing the endpoint titer by the IgA concentration of the sample. A subject with a  $\ge$ 4-fold increase in the specific IgA per total IgA content between pre- and any post-challenge specimens is considered an immunologic responder. All statistical analyses will be performed on  $\log_{10}$ -transformed titer values.

Salivary IgA: Total IgA content in the salivary extract samples will be determined by a modified ELISA method using commercial purified total IgA standard. Specimens with an IgA concentration  $<10 \mu g/mL$  will be excluded from all assessments of responder rates. Specific antibody levels in the salivary extracts will be determined using similar ELISA methods to those described above. Salivary antibodies will be reported as adjusted endpoint titers. A subject with a  $\ge$ 4-fold increase in the specific IgA per total IgA content between pre- and any post-challenge specimens is considered an immunologic responder. All statistical analyses will be performed on  $\log_{10}$ -transformed titer values.

In addition to the analyses detailed above, several post hoc analyses will be performed in an effort to further characterize the safety and immunogenicity of the study products. Estimated parameters not on the same scale as raw observations (e.g., regression coefficients) will be reported to 3 significant digits.

#### 11 General Statistical Considerations

All analyses will be grouped by cohort (1A, 1B, 2A, 2B). Generally, all data will be listed by cohort and subject. All summary tables will be structured with a column for each cohort and include an annotation for the total population size relevant to the table.

#### 12 Reporting Conventions

P-values ≥0.001 will be reported to 3 decimal places; p-values less than 0.001 will be reported as '<0.001'. Means, standard deviations, and any other statistics other than quantiles will be reported to one decimal place greater than the original data. Quantiles, such as median, or minimum and maximum will use the same number of decimal places.

#### 13 Technical Details

Statistical analyses will be performed using SAS v9.4 or newer for Windows (The SAS Institute, Cary, NC) and RStudio 2022.02.0 + 443 "Prairie Trillium" Release for Windows.

#### 14 Summary of Changes to Planned Analyses Outlined in Protocol

The analysis population definitions were modified from those originally outlined in the study protocol to better align with the planned study analyses.

#### 15 Appendices

#### 15.1 Sample Data Tables and Figures for Final Clinical Study Report

Sample data tables and figures to be included in the final clinical study report are included below to guide the analysis and data presentation. Final tables and figures may be modified to optimize data presentation.

Figures

Figure 1: Disposition of Subjects



#### **Listings**

**Listing 1: Demographics - Safety Population** 

| Subject ID | Sex | Race | Ethnicity | Age (years) |
|------------|-----|------|-----------|-------------|

21

Listing 2: Pre-Existing Medical Conditions - Safety Population

Listing 3: Solicited Adverse Events - Safety Population

| | Outcome | |
|---|---|---|
| | Relationship<br>to<br>Antibiotics | |
| | Severity Relationship to Challenge | |
| | Severity | |
| | End<br>Date | - |
| | Start<br>Date | |
| oparacon. | MedDRA®<br>Preferred<br>Term | |
| | MedDRA®<br>SOC | ٠,٠ |
| rishing of pointing fraction of the party of | AE<br>Description | |
| CONTRACTOR | Study<br>Group | |
| Simon | Subject Study<br>ID Group | 1 |

AE: adverse event; MedDRA®: Medical Dictionary for Regulatory Activities; SOC: system organ class

Tables with similar format to Listing 3:

Listing 4: Unsolicited Adverse Events - Safety Population

Listing 5: Serious Adverse Events - Safety Population

Listing 6: Vital Signs by Subject - Safety Population

| ) | • | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject ID Study Croun Study Day | Study Day | Doto | Time | Temperature | | Systolic BP | Systolic BP Diastolic BP |
| oun bect in | Study Group | Study Day | Date | 211112 | (°F) | (pbm) | (mm Hg) | (mm Hg) |
| , , , , , | | | | | | | | |

BP: blood pressure

| | Eosinophils | (cells/mm <sup>3</sup> ) |
|---|---|---|
| | <b>Platelets</b> | (cells/mm <sup>3</sup> ) |
| | Hemoglobin | (g/dL) |
| opulation | Leukocytes Neutrophils Lymphocytes Hemoglobin | |
| Values by Subject - Safety Population | Neutrophils | (cells/mm <sup>3</sup> ) (cells/mm <sup>3</sup> ) |
| | Leukocytes | (cells/mm <sup>3</sup> ) |
| Laboratory | Doto | Date |
| ematology | Study | Day |
| sting of He | Study | Group |
| Listing 7: Listing of Hematology Laboratory | Subject ID | Subjection |

Safety Population Listing 8: Listing of Chemistry Laboratory Values by Subject

| | Glucose | (mg/dL) |
|---|---|---|
| | BUN | (mg/dL) |
| | Potassium | (mEq/L) |
| | Sodium | (mEq/L) |
| aines by Subject - Saiety Fopulation | Creatinine | (mg/dL) |
| Dject - Saiet | $\mathbf{I}\mathbf{T}\mathbf{V}$ | (u/L) |
| values by Su | <b>LSV</b> | (n/L) |
| aboratory | Doto | Date |
| emistry La | Study | Day |
| Sting of Cr | Study | Group |
| LISTING 6: LISTING OF CHEMISTRY LABORATORY V | Subject ID | an palanc |

22

Listing 9: Listing of Concomitant Medications by Subject - Safety Population

| | Indication | | | | |
|---|---|---|---|---|---|
| | Date<br>Stopped | | | | |
| | Date<br>Started | | | | |
| | Route | | | | |
| ey i opanano | Frequency | | | | |
| abject - Sare | Unit | | | | |
| nearrouns by E | Dose | | | | |
| VIIII TALVA | Medication | | | | |
| disting / this and of concomment introductions by subject party to paradon | Study<br>Group | | | | |
| manue /· ma | Subject ID | | | | |
| | _ | - | - | - | <br>- |

Listing 10: Listing of Subject-Specific Protocol Deviations - Safety Population

| | | | 2 | | | | | , |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Study Crouns | Doto | Protocol | Reason for | Resulted in | Deviation | Deviation | |
| | dno o dnos | Date | Deviation | Deviation | AE | Category | Resolution | |
| | | | | | | | | _ |
| | | | • | | • | | | 1 |

AE: adverse event

| | Deviation<br>Resolution |
|---|---|
| | Deviation Category |
| Safety Population | Resulted in AE |
| c Protocol Deviations - Safety Population | Reason for<br>Deviation |
| Non-Subject-Specific | Protocol Deviation |
| Listing 11: Listing of Non-Subject-Specifi | Date |

AE: adverse event

Listing 12: Subjects Withdrawn or Lost to Follow-Up - Safety Population

| Subject ID Date of Last Visit Reason for Withdrawal/Loss to Follow-Up |
|---|
| <br>Date of Last Visit |
| <br>Subject ID |

Listing 13: Stool Log Listing - Safety Population

| 1 | 1 |
|-----------|---------------------|
| | Culture<br>Result |
| | Gross Blood Present |
| | Weight (g) |
| | Grade |
| | Collection<br>Time |
| | Collection<br>Date |
| | Study Day |
| J C 8 8 8 | Study<br>Group |
| | Subject ID |

Listing 14: Challenge Administration - Safety Population

| Time<br>Challenge<br>Administered |
|-----------------------------------|
| Time Buffer<br>Administered |
| Confirmed<br>Dose<br>(cfu) |
| Dose Prep<br>Time |
| Dose Date |
| Challenge<br>Strain |
| Study Group |
| Subject ID |

# Data Tables

Table 1: Demographics and Baseline Characteristics by Treatment Group - All Enrolled Subjects

| Table 1: Demographics and Dascinic Characteristics by Treatment Group - An Enronca Subjects | i actei istics n | y Heatinen | v - dnoin i | | unjeers | | |
|---|---|---|---|---|---|---|---|
| | lacksquare | Group 1B,<br>Naïve | Group 1B,<br>Veteran | Group 2A | Group 2B,<br>Naïve | Group 2B,<br>Veteran | All<br>Subjects |
| | (N=N) | (N=X) | (N=X) | (N=X) | | (N=X) | (N=X) |
| Sex [n (%)] | | | | | | | |
| Male | | | | | | | |
| Female | | | | | | | |
| Ethnicity [n (%)] | | | | | | | |
| Not Hispanic or Latino | | | | | | | |
| Hispanic or Latino | | | | | | | |
| Not Reported | | | | | | | |
| Unknown | | | | | | | |
| Race [n (%)] | | | | | | | |
| American Indian or Alaska Native | | | | | | | |
| Asian | | | | | | | |
| Native Hawaiian or Other Pacific Islander | | | | | | | |
| Black or African American | | | | | | | |
| White | | | | | | | |
| Multi-Racial | | | | | | | |
| Unknown | | | | | | | |
| Age (years) | | | | | | | |
| Mean (SD) | | | | | | | |
| Median | | | | | | | |
| Min/Max | | | | | | | |

SD: standard deviation

Table 2: Ineligibility Summary of Screen Failures

| nn n¹ |
|-------------------------------|
| Inclusion/Exclusion Criterion |
| Inclusion/Exclusion Category |

<sup>1</sup> More than one criterion may be marked per subject.

Table 3: Concomitant Medications by WHO Drug Classification - Safety Population [n (%)]

| Anatomical<br>Therapeutic | Medication Name | $\begin{bmatrix} \text{Group 1A} & (\text{N=X}) \end{bmatrix}$ | Group 1B,<br>Naïve | Group 1B, Group 1B, Naïve Veteran | Group 2A<br>(N=X) | Group 2B, Group 2B, Naïve Veteran | Group 2B,<br>Veteran | All<br>Subjects |
|---|---|---|---|---|---|---|---|---|
| Chemical | | | (N=X) | (N=X) | ` | $\overline{}$ | (N=X) | |
| [ATC 1] | [Medication 1] | | | | | | | |
| | [Medication 2] | | | | | | | |
| | [Medication 3] | | | | | | | |
| [ATC 2] | [Medication 1] | | | | | | | |
| | [Medication 2] | | | | | | | |
| | [Medication 3] | | | | | | | |

Table 4: Pre-Existing Medical Conditions by Treatment Group - Safety Population [n (%)]

| | | _ |
|---|---|---|
| | All Subjects<br>(N=X) | |
| | Group 2B, Veteran (N=X) | |
| [(a/)] | Group 2B,<br>Naïve<br>(N=X) | |
| morando - faci | Group 2A (N=X) | |
| ac drong | Group 1B,<br>Veteran<br>(N=X) | |
| | Group 1B,<br>Naïve<br>(N=X) | |
| out of the court | Group 1A<br>(N=X) | |
| (a) In manufactured and a summand of the manufactured and a summand of the manufactured and the summand of the | Medical Condition | |

Table 5: Adverse Events by MedDRA® System Organ Class (SOC), Preferred Term (PT), and Treatment Group Coded as 'Related' to Challenge - Safety Population [n (%)]

| System Organ Preferred Term Group 1A (N=X) Group 1B, Group 1B, (N=X) Group 2B, Naïve (N=X) Group 2B, Naïve (N=X) Group 2B, Naïve (N=X) All Subjects P-Value* [SOC 1] [PT 2] (N=X) (N=X) (N=X) (N=X) (N=X) (N=X) [SOC 1] [PT 2] (N=X) (N=X) (N=X) (N=X) (N=X) [SOC 2] [PT 3] (N=X) (N=X) (N=X) (N=X) (N=X) [SOC 2] [PT 2] (N=X) (N=X) (N=X) (N=X) (N=X) [SOC 2] [PT 2] (N=X) (N=X) (N=X) (N=X) (N=X) [SOC 2] [PT 2] (N=X) (N=X) (N=X) (N=X) (N=X) | | a Summan and | ndo - fam | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term (N=X) ( | System Organ | | Group 14 | Group 1B, | Group 1B, | Group 2A | Group 2B, | Group 2B, |
| [PT 1] (N=X) (N=X) (N=X) (N=X) (N=X) [PT 2] [PT 3] (N=X) (N=X) (N=X) [PT 2] [PT 1] (N=X) (N=X) (N=X) [PT 2] [PT 2] (N=X) (N=X) (N=X) [PT 2] [PT 3] (N=X) (N=X) (N=X) | Closs | Preferred Term | | Naïve | Veteran | N-N | Naïve | Veteran |
| | Class | | | (N=X) | (N=X) | (V_V) | (N=X) | (N=X) |
| | [SOC 1] | [PT 1] | | | | | | |
| | | [PT 2] | | | | | | |
| | | [PT 3] | | | | | | |
| [PT2] [PT3] | [SOC 2] | [PT 1] | | | | | | |
| [PT 3] | | [PT 2] | | | | | | |
| | | [PT 3] | | | | | | |

<sup>\*</sup>Between-group comparisons completed using Chi-squared analyses.

Table with similar format to Table 5:

Table 6: Adverse Events by MedDRA® System Organ Class (SOC), Preferred Term (PT), and Treatment Group Coded as 'Unrelated' to Challenge - Safety Population [n (%)]

Table 7: Severity of Solicited and Anticipated Adverse Events (Group 1A) - Per-Protocol Population [n (%)]

| | _ | | | ıp 1A<br>=X) | | |
|---|---|---|---|---|---|---|
| | None | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Total |
| Abdominal Cramps/Pain | | | | | | |
| Anorexia | | | | | | |
| Arthralgia | | | | | | |
| Bloating | | | | | | |
| Chills | | | | | | |
| Constipation | | | | | | |
| Flatulence | | | | | | |
| Myalgia | | | | | | |
| Headache | | | | | | |
| Lightheadedness | | | | | | |
| Malaise | | | | | | |
| Nausea | | | | | | |
| Tenesmus | | | | | | |
| Urgency | | | | | | |
| Diarrhea | | | | | | |
| Dysentery | | | | | | |
| Hypovolemia | | | | | | · |
| Fever | | | | | | |
| Vomiting | | | | | | |

Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: potentially life-threatening

Table with similar format to Table 7:

Table 8: Severity of Solicited and Anticipated Adverse Events (Group 2A) - Per-Protocol Population [n (%)]

Version 1.0; 04OCT2023 28

Table 9: Severity of Solicited and Anticipated Adverse Events (Group 1B) - Per-Protocol Population [n (%)]

| | | | Group 1 | np 1B, Naïve | , | | | | Group 1B, Veteran | , Veteran | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | <b>"</b> | =X) | • | | • | • | (N=X) | (X) | • | |
| | None | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Total | None | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Total |
| Abdominal | | | | | | | | | | | | |
| Cramps/Pain | | | | | | | | | | | | |
| Anorexia | | | | | | | | | | | | |
| Arthralgia | | | | | | | | | | | | |
| Bloating | | | | | | | | | | | | |
| Chills | | | | | | | | | | | | |
| Constipation | | | | | | | | | | | | |
| Flatulence | | | | | | | | | | | | |
| Myalgia | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | |
| Lightheadedness | | | | | | | | | | | | |
| Malaise | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | |
| Tenesmus | | | | | | | | | | | | |
| Urgency | | | | | | | | | | | | |
| Diarrhea | | | | | | | | | | | | |
| Dysentery | | | | | | | | | | | | |
| Hypovolemia | | | | | | | | | | | | |
| Fever | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | |
| Cundo 1, mildi Cundo J. modowata, Cundo 2, garrano | 7. modern | 10. Condo 2. 0 | | 1 | 1. 1. 2. 4. 2. 4. 1. | | | | | | | • |

Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: potentially life-threatening

Table with similar format to Table 9:

Table 10: Severity of Solicited and Anticipated Adverse Events (Group 2B) - Per-Protocol Population [n (%)]

Table 11: Rates of Shigellosis (95% CI) and Constitutional/Enteric Symptoms Following Shigella Challenge - Per-Protocol

| Population | , | | • | • | ) | ) | |
|---|---|---|---|---|---|---|---|
| | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B,<br>Veteran<br>(N=X) | Group 2A<br>(N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B,<br>Veteran<br>(N=X) | All Subjects (N=X) |
| Shigellosis | | | | | | | |
| Any Diarrhea | | | | | | | |
| Mild Diarrhea | | | | | | | |
| Moderate Diarrhea | | | | | | | |
| Severe Diarrhea | | | | | | | |
| More Severe Diarrhea | | | | | | | |
| Dysentery | | | | | | | |
| Fever (any severity) | | | | | | | |
| Moderate/Severe Abdominal Pain/Cramps | | | | | | | |
| Moderate/Severe Nausea | | | | | | | |
| Moderate/Severe Vomiting | | | | | | | |
| Moderate/Severe Anorexia | | | | | | | |
| Moderate/Severe Myalgia | | | | | | | |
| Moderate/Severe Arthralgia | | | | | | | |
| Moderate/Severe Malaise | | | | | | | |

30

31

| | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B,<br>Veteran<br>(N=X) | Group 2A<br>(N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B,<br>Veteran<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Maximum number of | Mean | | | | | | | |
| loose stools in 24h | Median | | | | | | | |
| | SD | | | | | | | |
| | Range | | | | | | | |
| Maximum volume of | Mean | | | | | | | |
| loose stools in 24h (g) | Median | | | | | | | |
| | SD | | | | | | | |
| | Range | | | | | | | |
| Total number of loose | Mean | | | | | | | |
| stools | Median | | | | | | | |
| | SD | | | | | | | |
| | Range | | | | | | | |
| Total volume of loose | Mean | | | | | | | |
| stools (g) | Median | | | | | | | |
| | SD | | | | | | | |
| | Range | | | | | | | |
| Maximum temperature | Mean | | | | | | | |
| (°F) | Median | | | | | | | |
| | SD | | | | | | | |
| | Range | | | | | | | |
| Time to diarrhea onset | Mean | | | | | | | |
| | Median | | | | | | | |
| | SD | | | | | | | |
| | Range | | | | | | | |
| Time to first Shigella- | Mean | | | | | | | |
| positive stool | Median | | | | | | | |
| | SD | | | | | | | |

| | Statistic | Group 1A (N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Group 1B, Naïve Veteran (N=X) (N=X) | Group 2A (N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B, Veteran (N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|---|---|
| | Range | | | | | | | |
| Shigella clinical severity | Mean | | | | | | | |
| score | Median | | | | | | | |
| | QS | | | | | | | |
| | Range | | | | | | | |

SD: standard deviation

#### 15.2 Sample Data Tables and Figures for Exploratory Analyses

Sample data tables and figures for exploratory analyses are included below to guide the analysis and data presentation. Final tables and figures may be modified to optimize data presentation.

#### **Listings**

Listing 15: Listing of Serologic IgG Responses to S. flexneri 2a Invaplex by Subject - Immunology Population

| Subject<br>ID | Study<br>Group | Baseline | Day 8 | Day 15 | Day 29 | Day 57 | <b>Day 90</b> | Day 180 |
|---|---|---|---|---|---|---|---|---|

Tables with similar format to Listing 15:

- Listing 16: Listing of Serologic IgA Responses to S. flexneri 2a Invaplex by Subject Immunology Population
- Listing 17: Listing of Serologic IgG Responses to *S. flexneri* 2a LPS by Subject Immunology Population
- Listing 18: Listing of Serologic IgA Responses to *S. flexneri* 2a LPS by Subject Immunology Population
- Listing 19: Listing of Serologic IgG Responses to *S. flexneri* 2a IpaB by Subject Immunology Population
- Listing 20: Listing of Serologic IgA Responses to S. flexneri 2a IpaB by Subject Immunology Population
- Listing 21: Listing of Serologic IgG Responses to S. flexneri 2a IpaC by Subject Immunology Population
- Listing 22: Listing of Serologic IgA Responses to S. flexneri 2a IpaC by Subject Immunology Population
- Listing 23: Listing of Serologic IgG Responses to S. flexneri 2a IpaD by Subject Immunology Population
- Listing 24: Listing of Serologic IgA Responses to *S. flexneri* 2a IpaD by Subject Immunology Population
- Listing 25: Listing of Serologic IgG Responses to S. sonnei Invaplex by Subject Immunology Population
- Listing 26: Listing of Serologic IgA Responses to *S. sonnei* Invaplex by Subject Immunology Population
- Listing 27: Listing of Serologic IgG Responses to S. sonnei LPS by Subject Immunology Population
- Listing 28: Listing of Serologic IgA Responses to S. sonnei LPS by Subject Immunology Population
- Listing 29: Listing of Serologic IgG Responses to S. sonnei IpaB by Subject Immunology Population

- Listing 30: Listing of Serologic IgA Responses to *S. sonnei* IpaB by Subject Immunology Population
- Listing 31: Listing of Serologic IgG Responses to *S. sonnei* IpaC by Subject Immunology Population
- Listing 32: Listing of Serologic IgA Responses to *S. sonnei* IpaC by Subject Immunology Population
- Listing 33: Listing of Serologic IgG Responses to S. sonnei IpaD by Subject Immunology Population
- Listing 34: Listing of Serologic IgA Responses to *S. sonnei* IpaD by Subject Immunology Population

Listing 35: Listing of Antibody in Lymphocyte Supernatant (ALS) IgG Responses to S. flexneri 2a Invaplex by Subject - Immunology Population

| Subject ID | Study Group | Baseline | Day 4 | Day 6 | Day 8 |
|------------|-------------|----------|-------|-------|-------|

Tables with similar format to Listing 35:

- Listing 36: Listing of ALS IgA Responses to S. flexneri 2a Invaplex by Subject Immunology Population
- Listing 37: Listing of ALS IgG Responses to *S. flexneri* 2a LPS by Subject Immunology Population
- Listing 38: Listing of ALS IgA Responses to *S. flexneri* 2a LPS by Subject Immunology Population
- Listing 39: Listing of ALS IgG Responses to *S. flexneri* 2a IpaB by Subject Immunology Population
- Listing 40: Listing of ALS IgA Responses to *S. flexneri* 2a IpaB by Subject Immunology Population
- Listing 41: Listing of ALS IgG Responses to *S. flexneri* 2a IpaC by Subject Immunology Population
- Listing 42: Listing of ALS IgA Responses to *S. flexneri* 2a IpaC by Subject Immunology Population
- Listing 43: Listing of ALS IgG Responses to *S. flexneri* 2a IpaD by Subject Immunology Population
- Listing 44: Listing of ALS IgA Responses to *S. flexneri* 2a IpaD by Subject Immunology Population
- Listing 45: Listing of ALS IgG Responses to *S. sonnei* Invaplex by Subject Immunology Population
- Listing 46: Listing of ALS IgA Responses to *S. sonnei* Invaplex by Subject Immunology Population
- Listing 47: Listing of ALS IgG Responses to S. sonnei LPS by Subject Immunology Population
- Listing 48: Listing of ALS IgA Responses to S. sonnei LPS by Subject Immunology Population
- Listing 49: Listing of ALS IgG Responses to S. sonnei IpaB by Subject Immunology Population
- Listing 50: Listing of ALS IgA Responses to S. sonnei IpaB by Subject Immunology Population
- Listing 51: Listing of ALS IgG Responses to *S. sonnei* IpaC by Subject Immunology Population
- Listing 52: Listing of ALS IgA Responses to *S. sonnei* IpaC by Subject Immunology Population
- Listing 53: Listing of ALS IgG Responses to *S. sonnei* IpaD by Subject Immunology Population
- Listing 54: Listing of ALS IgA Responses to *S. sonnei* IpaD by Subject Immunology Population

Listing 55: Listing of Fecal IgA Responses to S. flexneri 2a Invaplex by Subject - Immunology Population

| Subject ID | Study Group | Baseline | Day 4 | Day 8 | Day 15 | Day 29 |
|------------|-------------|----------|-------|-------|--------|--------|

Tables with similar format to Listing 55:

- Listing 56: Listing of Fecal IgA Responses to *S. flexneri* 2a LPS by Subject Immunology Population
- Listing 57: Listing of Fecal IgA Responses to *S. flexneri* 2a IpaB by Subject Immunology Population
- Listing 58: Listing of Fecal IgA Responses to *S. flexneri* 2a IpaC by Subject Immunology Population
- Listing 59: Listing of Fecal IgA Responses to *S. flexneri* 2a IpaD by Subject Immunology Population
- Listing 60: Listing of Fecal IgA Responses to S. sonnei Invaplex by Subject Immunology Population
- Listing 61: Listing of Fecal IgA Responses to *S. sonnei* LPS by Subject Immunology Population
- Listing 62: Listing of Fecal IgA Responses to *S. sonnei* IpaB by Subject Immunology Population
- Listing 63: Listing of Fecal IgA Responses to S. sonnei IpaC by Subject Immunology Population
- Listing 64: Listing of Fecal IgA Responses to *S. sonnei* IpaD by Subject Immunology Population

Listing 65: Salivary IgA Responses to *S. flexneri* 2a Invaplex, Listing of Values by Subject - Immunology Population

| Subject<br>ID | Study<br>Group | Baseline | Day 2 | Day 4 | Day 6 | Day 8 | Day 15 | Day 29 | Day 57 |
|---|---|---|---|---|---|---|---|---|---|

Tables with similar format to - Immunology Population

### Listing 65:

- Listing 66: Listing of Salivary IgA Responses to S. flexneri 2a LPS by Subject Immunology Population
- Listing 67: Listing of Salivary IgA Responses to S. flexneri 2a IpaB by Subject Immunology Population
- Listing 68: Listing of Salivary IgA Responses to S. flexneri 2a IpaC by Subject Immunology Population
- Listing 69: Listing of Salivary IgA Responses to S. flexneri 2a IpaD by Subject Immunology Population
- Listing 70: Listing of Salivary IgA Responses to *S. sonnei* Invaplex by Subject Immunology Population
- Listing 71: Listing of Salivary IgA Responses to *S. sonnei* LPS by Subject Immunology Population
- Listing 72: Listing of Salivary IgA Responses to *S. sonnei* IpaB by Subject Immunology Population
- Listing 73: Listing of Salivary IgA Responses to S. sonnei IpaC by Subject Immunology Population
- Listing 74: Listing of Salivary IgA Responses to S. sonnei IpaD by Subject Immunology Population

Data Tables

Table 13: Number of Immunology Samples Collected and Analyzed (Group 1A)<sup>1</sup> - Immunology Population

| Assay | Baseline <sup>2</sup> | Day 2 | Day 4 | Day 6 | Day 8 | <b>Day 15</b> | Day 29 | Day 57 | Day 90 | Day 180 |
|---|---|---|---|---|---|---|---|---|---|---|
| Serology | | | | | | | | | | |
| S. flexneri 2a Invaplex IgA | | | | | | | | | | |
| S. flexneri 2a Invaplex IgG | | | | | | | | | | |
| S. flexneri 2a LPS IgA | | | | | | | | | | |
| S. flexneri 2a LPS IgG | | | | | | | | | | |
| S. flexneri 2a IpaB IgA | | | | | | | | | | |
| S. flexneri 2a IpaB IgG | | | | | | | | | | |
| S. flexneri 2a IpaC IgA | | | | | | | | | | |
| S. flexneri 2a IpaC IgG | | | | | | | | | | |
| S. flexneri 2a IpaD IgA | | | | | | | | | | |
| S. flexneri 2a IpaD IgG | | | | | | | | | | |
| S. sonnei Invaplex IgA | | | | | | | | | | |
| S. sonnei Invaplex IgG | | | | | | | | | | |
| S. sonnei LPS IgA | | | | | | | | | | |
| S. sonnei LPS IgG | | | | | | | | | | |
| S. sonnei IpaB IgA | | | | | | | | | | |
| S. sonnei IpaB IgG | | | | | | | | | | |
| S. sonnei IpaC IgG | | | | | | | | | | |
| S. sonnei IpaC IgA | | | | | | | | | | |
| S. sonnei IpaD IgA | | | | | | | | | | |
| S. sonnei IpaD IgG | | | | | | | | | | |
| ALS | | | | | | | | | | |
| S. flexneri 2a Invaplex IgA | | | | | | | | | | |
| S. flexneri 2a Invaplex IgG | | | | | | | | | | |
| S. flexneri 2a LPS IgA | | | | | | | | | | |
| S. flexneri 2a LPS IgG | | | | | | | | | | |
| S. flexneri 2a IpaB IgA | | | | | | | | | | |

| Assay | Baseline <sup>2</sup> | Day 2 | Day 4 | Day 6 | Day 8 | Day 15 | Day 29 | <b>Day 57</b> | <b>Day 90</b> | Day 180 |
|---|---|---|---|---|---|---|---|---|---|---|
| S. flexneri 2a IpaB IgG | | | | | | | | | | |
| S. flexneri 2a IpaC IgA | | | | | | | | | | |
| S. flexneri 2a IpaC IgG | | | | | | | | | | |
| S. flexneri 2a IpaD IgA | | | | | | | | | | |
| S. flexneri 2a IpaD IgG | | | | | | | | | | |
| S. sonnei Invaplex IgA | | | | | | | | | | |
| S. sonnei Invaplex IgG | | | | | | | | | | |
| S. sonnei LPS IgA | | | | | | | | | | |
| S. sonnei LPS IgG | | | | | | | | | | |
| S. sonnei IpaB IgA | | | | | | | | | | |
| S. sonnei IpaB IgG | | | | | | | | | | |
| S. sonnei IpaC IgG | | | | | | | | | | |
| S. sonnei IpaC IgA | | | | | | | | | | |
| S. sonnei IpaD IgA | | | | | | | | | | |
| S. sonnei IpaD IgG | | | | | | | | | | |
| Fecal | | | | | | | | | | |
| S. flexneri 2a Invaplex IgA | | | | | | | | | | |
| S. flexneri 2a LPS IgA | | | | | | | | | | |
| S. flexneri 2a IpaB IgA | | | | | | | | | | |
| S. flexneri 2a IpaC IgA | | | | | | | | | | |
| S. flexneri 2a IpaD IgA | | | | | | | | | | |
| S. sonnei Invaplex IgA | | | | | | | | | | |
| S. sonnei LPS IgA | | | | | | | | | | |
| S. sonnei IpaB IgA | | | | | | | | | | |
| S. sonnei IpaC IgA | | | | | | | | | | |
| S. sonnei IpaD IgA | | | | | | | | | | |
| Salivary | | | | | | | | | | |
| S. flexneri 2a Invaplex IgA | | | | | | | | | | |
| S. flexneri 2a LPS IgA | | | | | | | | | | |
| S. flexneri 2a IpaB IgA | | | | | | | | | | |

| Assay | Baseline <sup>2</sup> Day 2 | Day 2 | Day 4 | Day 6 | Day 8 | Day 8 Day 15 | Day 29 | Day 57 | Day 90 | Day 180 |
|---|---|---|---|---|---|---|---|---|---|---|
| S. flexneri 2a IpaC IgA | | | | | | | | | | |
| S. flexneri 2a IpaD IgA | | | | | | | | | | |
| S. sonnei Invaplex IgA | | | | | | | | | | |
| S. sonnei LPS IgA | | | | | | | | | | |
| S. sonnei IpaB IgA | | | | | | | | | | |
| S. sonnei IpaC IgA | | | | | | | | | | |
| S. sonnei IpaD IgA | | | | | | | | | | |

Analyzed by the lab and data available.

IgA: immunoglobulin A; IgG: immunoglobulin G; LPS: Iipopolysaccharide; IpaB: invasin plasmid antigen B; IpaC: invasin plasmid antigen C; IpaD: invasin plasmid antigen D; ALS: antibody in lymphocyte supernatant

## Tables with similar format to Table 13:

Table 15: Number of Immunology Samples Collected and Analyzed (Group 2A) - Immunology Population Table 14: Number of Immunology Samples Collected and Analyzed (Group 1B) - Immunology Population Table 16: Number of Immunology Samples Collected and Analyzed (Group 2B) - Immunology Population

<sup>&</sup>lt;sup>2</sup> Most recent observation prior to challenge.

44

Table 17: Serologic IgG Responses to S. flexneri 2a Invaplex, Descriptive Statistics by Study Day and Study Group -Immunology Population\*

| Group 1B, Group 2A Group 2B, Veteran (N=X) (N=X) (N=X) (N=X) (N=X) | | Ov 1 | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Mean xxx.x Median xxx.x SD xxx.x Xxx.x Xxx.x< | Time Point | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Veteran (N=X) | Group 2A (N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B, Veteran (N=X) |
| Mean xxx SD xxx Range xxxxx, n Mean Median Nean n Median SD Range n Median SD Range n Median Median Median SD Median SD Range Range Nean Range Range Range Range | Baseline | n | XX | | | | | |
| Median xxx SD xxxx, Range xxxxx, n Median SD Range n Median Nange n Median n Range n Median n Median Median SD Range SD Range Range Range Range Range | | Mean | XXXX.X | | | | | |
| SD xxx Range xxxx, n Mean Median Nedian SD Range n Median Nange Nedian Nange Nedian Nedian Nedian Median Nedian SD Range Range Nedian SD Range Range Range | | Median | XXXX | | | | | |
| Range xxxx, n Mean Median Median SD Median Range n Median m Median m Median m Median Median SD Median SD Median SD Median SD Median SD Range Range m Range m Range m Range m | | SD | XXX.X | | | | | |
| | | Range | XXXX, XXXX | | | | | |
| | Day 8 | и | | | | | | |
| | | Mean | | | | | | |
| | | Median | | | | | | |
| | | SD | | | | | | |
| | | Range | | | | | | |
| | Day 15 | u | | | | | | |
| | | Mean | | | | | | |
| | | Median | | | | | | |
| | | SD | | | | | | |
| | | Range | | | | | | |
| | Day 29 | и | | | | | | |
| | | Mean | | | | | | |
| | | Median | | | | | | |
| | | SD | | | | | | |
| | | Range | | | | | | |
| Mean Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median Median <td>Day 57</td> <td>u</td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> | Day 57 | u | | | | | | |
| Median SD Range | | Mean | | | | | | |
| SD Range | | Median | | | | | | |
| Range | | SD | | | | | | |
| | | Range | | | | | | |

| ٧<br>/ | † |
|--------|---|

| | Time Point | Statistic | Group 1A (N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Veteran (N=X) | Group 2A<br>(N=X) | Group 2B, Naïve (N=X) | Group 2B, Veteran (N=X) |
|---|---|---|---|---|---|---|---|---|
| | Day 90 | u | | | | | | |
| | | Mean | | | | | | |
| | | Median | | | | | | |
| | | SD | | | | | | |
| | | Range | | | | | | |
| Mean Median Pange Range Range Range | Day 180 | n | | | | | | |
| Median SD Range | | Mean | | | | | | |
| SD Range Ra | | Median | | | | | | |
| Range | | SD | | | | | | |
| | | Range | | | | | | |

IgG: immunoglobulin G; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; SD: standard

Tables with similar format to Table 17:

 
 Table 18: Serologic IgA Responses to S. flexneri 2a Invaplex, Descriptive Statistics by Study Day and Study Group Immunology Population

Table 19: Serologic IgG Responses to S. flexneri 2a LPS, Descriptive Statistics by Study Day and Study Group -Immunology Population

Table 20: Serologic IgA Responses to S. flexneri 2a LPS, Descriptive Statistics by Study Day and Study Group -Immunology Population

Table 21: Serologic IgG Responses to S. flexneri 2a IpaB, Descriptive Statistics by Study Day and Study Group -Immunology Population

Table 22: Serologic IgA Responses to S. flexneri 2a IpaB, Descriptive Statistics by Study Day and Study Group Immunology Population Table 23: Serologic IgG Responses to S. flexneri 2a IpaC, Descriptive Statistics by Study Day and Study Group -Immunology Population

<sup>\*</sup>Log10 titers used to summarize these data.

- Table 24: Serologic IgA Responses to S. flexneri 2a IpaC, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 25: Serologic IgG Responses to S. flexneri 2a IpaD, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 26: Serologic IgA Responses to S. flexneri 2a IpaD, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 27: Serologic IgG Responses to S. sonnei Invaplex, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 28: Serologic IgA Responses to S. sonnei Invaplex, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 29: Serologic IgG Responses to S. sonnei LPS, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 30: Serologic IgA Responses to S. sonnei LPS, Descriptive Statistics by Study Day and Study Group -
  - Table 31: Serologic IgG Responses to S. sonnei IpaB, Descriptive Statistics by Study Day and Study Group -Immunology Population Immunology Population
- Serologic IgA Responses to S. sonnei IpaB, Descriptive Statistics by Study Day and Study Group Immunology Population
  - Table 33: Serologic IgG Responses to S. sonnei IpaC, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 34: Serologic IgA Responses to S. sonnei IpaC, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 35: Serologic IgG Responses to S. sonnei IpaD, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 36: Serologic IgA Responses to S. sonnei IpaD, Descriptive Statistics by Study Day and Study Group -**Immunology Population**

Table 37: Antibody in Lymphocyte Supernatant (ALS) IgG Responses to S. flexneri 2a Invaplex, Descriptive Statistics by Study Day and Study Group - Immunology Population\*

| Time Point | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Veteran (N=X) | Group 2A<br>(N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B, Veteran (N=X) |
|---|---|---|---|---|---|---|---|
| Baseline | n | XX | | | | | |
| | Mean | XXXX.X | | | | | |
| | Median | XXXX | | | | | |
| | SD | XXXX.X | | | | | |
| | Range | XXXX, XXXX | | | | | |
| Day 4 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 6 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 8 | и | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| 1. J. | I. O. imana and benefit O. M. mana and a survey in | | 0.40[ | the immense and it is a completion or another of which date at the consist of the standard | oft to stale driver aton | | CD. standand |

IgG: immunoglobulin G; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; SD: standard deviation

<sup>\*</sup>Log10 titers used to summarize these data.

### Tables with similar format to Table 37:

- Table 38: ALS IgA Responses to S. flexneri 2a Invaplex, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 39: ALS IgG Responses to S. flexneri 2a LPS, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 40: ALS IgA Responses to S. flexneri 2a LPS, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 41: ALS IgG Responses to S. flexneri 2a IpaB, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 42: ALS IgA Responses to S. flexneri 2a IpaB, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 43: ALS IgG Responses to S. flexneri 2a IpaC, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 44: ALS IgA Responses to S. flexneri 2a IpaC, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 45: ALS IgG Responses to S. flexneri 2a IpaD, Descriptive Statistics by Study Day and Study Group -**Immunology Population**
- Table 46: ALS IgA Responses to S. flexneri 2a IpaD, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 47: ALS IgG Responses to S. sonnei Invaplex, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 48: ALS IgA Responses to S. sonnei Invaplex, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 49: ALS IgG Responses to S. sonnei LPS, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 50: ALS IgA Responses to S. sonnei LPS, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 51: ALS IgG Responses to S. sonnei IpaB, Descriptive Statistics by Study Day and Study Group Immunology Population

- Table 53: ALS IgG Responses to S. sonnei IpaC, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 54: ALS IgA Responses to S. sonnei IpaC, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 55: ALS IgG Responses to S. sonnei IpaD, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 56: ALS IgA Responses to S. sonnei IpaD, Descriptive Statistics by Study Day and Study Group Immunology Population

50

Table 57: Fecal IgA Responses to S. flexneri 2a Invaplex, Descriptive Statistics by Study Day and Study Group - Immunology Population\*

| Time Point | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Veteran (N=X) | Group 2A<br>(N=X) | Group 2B, Naïve (N=X) | Group 2B, Veteran (N=X) |
|---|---|---|---|---|---|---|---|
| Baseline | u | XX | | | | | |
| | Mean | XXX.X | | | | | |
| | Median | XXXX | | | | | |
| | SD | XXXX.X | | | | | |
| | Range | XXXX, XXXX | | | | | |
| Day 4 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 8 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 15 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 29 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |

IgA: immunoglobulin A; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; SD: standard

Tables with similar format to Table 57:

Table 58: Fecal IgA Responses to S. flexneri 2a LPS, Descriptive Statistics by Study Day and Study Group -Immunology Population Table 59: Fecal IgA Responses to S. flexneri 2a IpaB, Descriptive Statistics by Study Day and Study Group -Immunology Population Table 60: Fecal IgA Responses to S. flexneri 2a IpaC, Descriptive Statistics by Study Day and Study Group -**Immunology Population**  Table 61: Fecal IgA Responses to S. flexneri 2a IpaD, Descriptive Statistics by Study Day and Study Group -**Immunology Population**  Table 62: Fecal IgA Responses to S. sonnei Invaplex, Descriptive Statistics by Study Day and Study Group **Immunology Population**  Table 63: Fecal IgA Responses to S. sonnei LPS, Descriptive Statistics by Study Day and Study Group - Immunology Population Table 64: Fecal IgA Responses to S. sonnei IpaB, Descriptive Statistics by Study Day and Study Group - Immunology Population Table 65: Fecal IgA Responses to S. sonnei IpaC, Descriptive Statistics by Study Day and Study Group - Immunology Population

Table 66: Fecal IgA Responses to S. sonnei IpaD, Descriptive Statistics by Study Day and Study Group - Immunology Population

<sup>\*</sup>Log10 titers used to summarize these data.

52

Table 67: Salivary IgA Responses to S. flexneri 2a Invaplex, Descriptive Statistics by Study Day and Study Group -Immunology Population\*

| | 1 30 | ē | | | | | |
|---|---|---|---|---|---|---|---|
| Time Point | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Veteran (N=X) | Group 2A<br>(N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B, Veteran (N=X) |
| Baseline | n | XX | | | | | |
| | Mean | XXXX.X | | | | | |
| | Median | XXXX | | | | | |
| | SD | XXXX.X | | | | | |
| | Range | XXXX, XXXX | | | | | |
| Day 2 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 4 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 6 | n | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 8 | n | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 15 | n | | | | | | |

| Time Point | Statistic | Group 1A | Group 1B, | Group 1B,<br>Veteran | Group 2A | Group 2B, | Group 2B,<br>Veteran |
|---|---|---|---|---|---|---|---|
| | | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 29 | n | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |
| Day 57 | u | | | | | | |
| | Mean | | | | | | |
| | Median | | | | | | |
| | SD | | | | | | |
| | Range | | | | | | |

IgA: immunoglobulin A; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; SD: standard deviation

Tables with similar format to Table 67:

Table 68: Salivary IgA Responses to S. flexneri 2a LPS, Descriptive Statistics by Study Day and Study Group -Immunology Population Table 69: Salivary IgA Responses to S. flexneri 2a IpaB, Descriptive Statistics by Study Day and Study Group -Immunology Population

Table 70: Salivary IgA Responses to S. flexneri 2a IpaC, Descriptive Statistics by Study Day and Study Group -Immunology Population Table 71: Salivary IgA Responses to S. flexneri 2a IpaD, Descriptive Statistics by Study Day and Study Group -**Immunology Population** 

<sup>\*</sup>Log<sub>10</sub> titers used to summarize these data.

- Table 73: Salivary IgA Responses to S. sonnei LPS, Descriptive Statistics by Study Day and Study Group Immunology Population
- Table 74: Salivary IgA Responses to S. sonnei IpaB, Descriptive Statistics by Study Day and Study Group -Immunology Population
  - Table 75: Salivary IgA Responses to S. sonnei IpaC, Descriptive Statistics by Study Day and Study Group -Immunology Population
- Table 76: Salivary IgA Responses to S. sonnei IpaD, Descriptive Statistics by Study Day and Study Group -Immunology Population

55

Table 77: Serologic Responses to S. flexneri 2a Invaplex, Geometric Mean Titer by Study Day and Study Group - Immunology Population

| • | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B,<br>Veteran<br>(N=X) | Group 2A (N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B, Veteran (N=X) | P-Value1 |
| Serum IgA | | | , | | | , | , | |
| Baseline | n | XX | | | | | | |
| | GMT | XXXX | | | | | | X.XXXX |
| | 95% CI | XXXX, XXXX | | | | | | |
| Day 8 | n | XX | | | | | | |
| | GMT | XXXX | | | | | | |
| | 95% CI | XXXX, XXXX | | | | | | |
| | GMFR | XXXX | | | | | | |
| | <b>GMFR 95% CI</b> | XXXX, XXXX | | | | | | |
| Day 15 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 29 | n | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 57 | n | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 90 | n | | | | | | | |

| Time Doint | Statistic | Group 1A | Group 1B, | Group 1B, | Group 2A | Group 2B, | Group 2B, | D Volue |
|---|---|---|---|---|---|---|---|---|
| | Statistic | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | ı -v anuc |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 180 | n | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Serum IgG | | | | | | | | |
| Baseline | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| Day 8 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |
| Day 15 | n | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |
| Day 29 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |

| $\Gamma$ |
|----------|
| 1 |
| • |

| Ē | | Group 1A | Group 1B, | Group 1B, | Group 2A | Group 2B, | Group 2B, | 1 V V J |
|---|---|---|---|---|---|---|---|---|
| Time Foint | Statistic | (N=N) | Naive<br>(N=X) | v eteran<br>(N=X) | (N=X) | (N=X) | v eteran<br>(N=X) | r-v aiue: |
| Day 57 | n | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |
| Day 90 | n | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 180 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |

IgA: immunoglobulin A; IgG: immunoglobulin G; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; GMT: geometric mean titer; CI: confidence interval; GMFR: geometric mean fold-rise from baseline

Tables with similar format to Table 77:

Table 78: Serologic Responses to S. flexneri 2a LPS, Geometric Mean Titer by Study Day and Study Group -Immunology Population Table 79: Serologic Responses to S. flexneri 2a IpaB, Geometric Mean Titer by Study Day and Study Group -Immunology Population

Table 80: Serologic Responses to S. flexneri 2a IpaC, Geometric Mean Titer by Study Day and Study Group -Immunology Population Table 81: Serologic Responses to S. flexneri 2a IpaD, Geometric Mean Titer by Study Day and Study Group -Immunology Population

<sup>&#</sup>x27;P-values are from ANOVA tests of differences between groups in mean log titers.

- Table 83: Serologic Responses to S. sonnei LPS, Geometric Mean Titer by Study Day and Study Group Immunology Population
- Table 84: Serologic Responses to S. sonnei IpaB, Geometric Mean Titer by Study Day and Study Group Immunology

Population

- Table 85: Serologic Responses to S. sonnei IpaC, Geometric Mean Titer by Study Day and Study Group Immunology Population
- Table 86: Serologic Responses to S. sonnei IpaD, Geometric Mean Titer by Study Day and Study Group Immunology Population

59

Table 87: ALS Responses to S. flexneri 2a Invaplex, Geometric Mean Titer by Study Day and Study Group - Immunology Population

| tic (N=X) (N=X) (N=X) (N=X) xx xx xx xx xx xx xxx xxx | | | Cuom 1 | Group 1B, | Group 1B, | Cuomo 2 A | Group 2B, | Group 2B, | |
|---|---|---|---|---|---|---|---|---|---|
| BeA ne n GMT 95% CI GMFR | Time Point | Statistic | (N=X) | Naïve<br>(N=X) | Veteran<br>(N=X) | (N=X) | Naïve<br>(N=X) | Veteran<br>(N=X) | P-Value <sup>1</sup> |
| December | ALS IgA | | | | | | | | |
| GMT n GMT 95% CI GMT 95% CI GMFR GMFR 95% CI 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | Baseline | u | XX | | | | | | |
| 95% CI n GMT 95% CI GMFR GMFR 95% CI GMFR | | GMT | XXXX | | | | | | X.XXXX |
| n GMT 95% CI GMFR GMFR | | 95% CI | XXXX, XXXX | | | | | | |
| GMT 95% CI GMFR GMFR GMT 95% CI GMT 95% CI GMFR D O O O O O O O O O O O O | Day 4 | u | XX | | | | | | |
| 95% CI GMFR GMFR 95% CI n GMT 95% CI GMFR | | GMT | XXXX | | | | | | |
| GMFR 95% CI | | 95% CI | XXXX, XXXX | | | | | | |
| GMFR 95% CI | | GMFR | XXXX | | | | | | |
| D <sub>B</sub> au | | GMFR 95% CI | XXXX, XXXX | | | | | | |
| ည္အေျ | Day 6 | u | | | | | | | |
| ည္အ ချ | | GMT | | | | | | | |
| So e | | 95% CI | | | | | | | |
| ပ္တံ့ ခု | | GMFR | | | | | | | |
| Se en | | GMFR 95% CI | | | | | | | |
| <b>5</b> 9 9 | Day 8 | n | | | | | | | |
| Se e | | GMT | | | | | | | |
| Sg eu | | 95% CI | | | | | | | |
| <b>5</b> 8 | | GMFR | | | | | | | |
| Sg eu | | GMFR 95% CI | | | | | | | |
| eu | ALS IgG | | | | | | | | |
| | Baseline | u | | | | | | | |
| | | GMT | | | | | | | |
| | | 95% CI | | | | | | | |
| | Day 4 | п | | | | | | | |
| GMT | | GMT | | | | | | | |

| Time Point | Statistic | Group 1A | Group 1B,<br>Naïve | Group 1B,<br>Veteran | Group 2A | Group 2B,<br>Naïve | Group 2B,<br>Veteran | P-Value <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|
| | | (X=N) | (N=X) | (N=X) | (X=N) | (N=X) | (N=X) | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 6 | и | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |
| Day 8 | и | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |

number of subjects with data at the specified time point; GMT: geometric mean titer; CI: confidence interval; GMFR: geometric mean fold-rise from baseline ALS: antibody in lymphocyte supernatant; IgA: immunoglobulin A; IgG: immunoglobulin G; N: number of subjects in the immunogenicity population; n: P-values are from ANOVA tests of differences between groups in mean log titers.

Tables with similar format to Table 87:

 
 Fable 88: ALS Responses to S. flexneri 2a LPS, Geometric Mean Titer by Study Day and Study Group - Immunology
 Population Table 89: ALS Responses to S. flexneri 2a IpaB, Geometric Mean Titer by Study Day and Study Group - Immunology Population

Table 90: ALS Responses to S. flexneri 2a IpaC, Geometric Mean Titer by Study Day and Study Group - Immunology Population Table 91: ALS Responses to S. flexneri 2a IpaD, Geometric Mean Titer by Study Day and Study Group - Immunology Population

Table 92: ALS Responses to S. sonnei Invaplex, Geometric Mean Titer by Study Day and Study Group - Immunology Population

Version 1.0; 04OCT2023

- Table 94: ALS Responses to S. sonnei IpaB, Geometric Mean Titer by Study Day and Study Group Immunology Population
- Table 95: ALS Responses to S. sonnei IpaC, Geometric Mean Titer by Study Day and Study Group Immunology Population
- Table 96: ALS Responses to S. sonnei IpaD, Geometric Mean Titer by Study Day and Study Group Immunology Population

Table 97: Fecal IgA Responses to S. flexneri 2a Invaplex, Geometric Mean Titer by Study Day and Study Group -Immunology Population

| | minances repairment | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Group 14 | Group 1B, | Group 1B, | Group 24 | Group 2B, | Group 2B, | |
| Time Point | Statistic | (N=X) | Naïve<br>(N=X) | Veteran<br>(N=X) | (X=N) | Naïve<br>(N=X) | Veteran<br>(N=X) | P-Value <sup>1</sup> |
| Baseline | n | XX | | | | | | |
| | GMT | XXXX | | | | | | X.XXXX |
| | 95% CI | XXXX, XXXX | | | | | | |
| Day 4 | u | XX | | | | | | |
| | GMT | XXXX | | | | | | |
| | 95% CI | XXXX, XXXX | | | | | | |
| | GMFR | XXXX | | | | | | |
| | <b>GMFR 95% CI</b> | XXXX, XXXX | | | | | | |
| Day 8 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 15 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 29 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |
| Joloonimmi A T | and the stockers to me decree 1 1. A willing to account to | social contractions | in the contract of the contrac | | Af antigota with de | 1 2 2 th 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | mountain of anti- ante writh date at the an one that time as int. and | |

IgA: immunoglobulin A; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; GMT: geometric mean titer; CI: confidence interval; GMFR: geometric mean fold-rise from baseline

Version 1.0; 04OCT2023

- Tables with similar format to Table 97:
- Table 98: Fecal IgA Responses to S. flexneri 2a LPS, Geometric Mean Titer by Study Day and Study Group -Immunology Population
- Table 99: Fecal IgA Responses to S. flexneri 2a IpaB, Geometric Mean Titer by Study Day and Study Group Immunology Population
- Table 100: Fecal IgA Responses to S. flexneri 2a IpaC, Geometric Mean Titer by Study Day and Study Group Immunology Population
- Table 101: Fecal IgA Responses to S. flexneri 2a IpaD, Geometric Mean Titer by Study Day and Study Group -Immunology Population
- Table 102: Fecal IgA Responses to S. sonnei Invaplex, Geometric Mean Titer by Study Day and Study Group -Immunology Population
- Table 103: Fecal IgA Responses to S. sonnei LPS, Geometric Mean Titer by Study Day and Study Group Immunology Population
- Table 104: Fecal IgA Responses to S. sonnei IpaB, Geometric Mean Titer by Study Day and Study Group -**Immunology Population**
- Table 105: Fecal IgA Responses to S. sonnei IpaC, Geometric Mean Titer by Study Day and Study Group -**Immunology Population**
- Table 106: Fecal IgA Responses to S. sonnei IpaD, Geometric Mean Titer by Study Day and Study Group -Immunology Population

Table 107: Salivary IgA Responses to S. flexneri 2a Invaplex, Geometric Mean Titer by Study Day and Study Group - Immunology Population

| | Tarama In - 18 annum | | • | | • | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | Group 1A | Group 1B,<br>Naïve | Group 1B,<br>Veteran | Group 2A | Group 2B,<br>Naïve | Group 2B,<br>Veteran | P-Value <sup>1</sup> |
| | | (v_v) | (N=X) | (N=X) | (N-A) | (N=X) | (N=X) | |
| Baseline | n | XX | | | | | | |
| | GMT | XXXX | | | | | | X.XXXX |
| | 95% CI | XXXX, XXXX | | | | | | |
| Day 2 | u | XX | | | | | | |
| | GMT | XXXX | | | | | | |
| | 95% CI | XXXX, XXXX | | | | | | |
| | GMFR | XXXX | | | | | | |
| | GMFR 95% CI | XXXX, XXXX | | | | | | |
| Day 4 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |
| Day 6 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 8 | n | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 15 | n | | | | | | | |
| | GMT | | | | | | | |

| Time Point | Statistic | Group 1A | Group 1B,<br>Naïve | Group 1B,<br>Veteran | Group 2A | Group 2B,<br>Naïve | Group 2B,<br>Veteran | P-Value <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|
| | | (N=X) | (N=X) | | | (N=X) | (N=X) | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |
| Day 29 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | <b>GMFR 95% CI</b> | | | | | | | |
| Day 57 | u | | | | | | | |
| | GMT | | | | | | | |
| | 95% CI | | | | | | | |
| | GMFR | | | | | | | |
| | GMFR 95% CI | | | | | | | |

IgA: immunoglobulin A; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; GMT: geometric mean titer; CI: confidence interval; GMFR: geometric mean fold-rise from baseline

Tables with similar format to Table 107:

 
 Fable 108: Salivary IgA Responses to S. flexneri 2a LPS, Geometric Mean Titer by Study Day and Study Group Immunology Population Table 109: Salivary IgA Responses to S. flexneri 2a IpaB, Geometric Mean Titer by Study Day and Study Group -Immunology Population

Table 110: Salivary IgA Responses to S. flexneri 2a IpaC, Geometric Mean Titer by Study Day and Study Group Immunology Population Table 111: Salivary IgA Responses to S. flexneri 2a IpaD, Geometric Mean Titer by Study Day and Study Group Immunology Population

Table 112: Salivary IgA Responses to S. sonnei Invaplex, Geometric Mean Titer by Study Day and Study Group -**Immunology Population**  Version 1.0; 04OCT2023

P-values are from ANOVA tests of differences between groups in mean log titers.

- Table 114: Salivary IgA Responses to S. sonnei IpaB, Geometric Mean Titer by Study Day and Study Group -Immunology Population
  - Table 115: Salivary IgA Responses to S. sonnei IpaC, Geometric Mean Titer by Study Day and Study Group -Immunology Population
- Table 116: Salivary IgA Responses to S. sonnei IpaD, Geometric Mean Titer by Study Day and Study Group -Immunology Population

29

Table 117: Serologic Responses to S. flexneri 2a Invaplex, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

| Time Point | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Veteran (N=X) | Group 2A<br>(N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B, Veteran (N=X) | P-Value <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|
| Serum IgA | | | | | | | | |
| Day 8 | u | XX | | | | | | |
| | Responder % | XX.X | | | | | | X.XXXX |
| | 95% CI | XX.X, XX.X | | | | | | |
| Day 15 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 29 | n | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 57 | n | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 90 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 180 | n | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Serum IgG | | | | | | | | |
| Day 8 | п | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 15 | n | | | | | | | |
| | Responder % | | | | | | | |

| | Group 1A | Group 1B, | Group 1B, | Group 2A | Group 2B, | Group 2B, $V_{oforon}$ | D Voluol |
|---|---|---|---|---|---|---|---|
| (N=X) | | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | I -v aiuc |

IgA: immunoglobulin A; IgG: immunoglobulin G; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; Responder defined as ≥4-fold increase in titer from baseline; CI: Exact Clopper-Pearson Confidence Interval

Tables with similar format to Table 117:

Table 118: Serologic Responses to S. flexneri 2a LPS, Immunologic Responder Rates by Study Day and Study Group -Immunology Population Table 119: Serologic Responses to S. flexneri 2a IpaB, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

 
 Table 120: Serologic Responses to S. flexneri 2a IpaC, Immunologic Responder Rates by Study Day and Study Group Immunology Population  
 Table 121: Serologic Responses to S. flexneri 2a IpaD, Immunologic Responder Rates by Study Day and Study Group **Immunology Population** 

Table 122: Serologic Responses to S. sonnei Invaplex, Immunologic Responder Rates by Study Day and Study Group -**Immunology Population** 

Version 1.0; 04OCT2023

P-values are from Fisher's exact 2-tailed tests of differences between groups in immunologic responder rates.

- Table 123: Serologic Responses to S. sonnei LPS, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 124: Serologic Responses to S. sonnei IpaB, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 125: Serologic Responses to S. sonnei IpaC, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 126: Serologic Responses to S. sonnei IpaD, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

Table 127: ALS Responses to S. flexneri 2a Invaplex, Immunologic Responder Rates by Study Day and Study Group -**Immunology Population** 

| | | ( | Group 1B, | Group 1B, | ( | Group 2B, | Group 2B, | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | Group IA<br>(N=X) | Naïve<br>(N=X) | Veteran<br>(N=X) | Group 2A<br>(N=X) | Naïve<br>(N=X) | Veteran<br>(N=X) | P-Value <sup>1</sup> |
| ALS IgA | | | | , | | | | |
| Day 4 | n | XX | | | | | | |
| | Responder % | XX.X | | | | | | X.XXXX |
| | 95% CI | XX.X, XX.X | | | | | | |
| Day 6 | п | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 8 | n | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| ALS IgG | | | | | | | | |
| Day 4 | и | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 6 | n | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 8 | и | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| . 1 1.7 5 1 4 | VI O | 1. 1 | 1-1-1-1 | - | AI to and the second | 1 - 1 - 1 | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |

number of subjects with data at the specified time point; Responder defined as ≥4-fold increase in titer from baseline; CI: Exact Clopper-Pearson Confidence ALS: antibody in lymphocyte supernatant; IgA: immunoglobulin A; IgG: immunoglobulin G; N: number of subjects in the immunogenicity population; n: Interval

<sup>&</sup>lt;sup>1</sup>P-values are from Fisher's exact 2-tailed tests of differences between groups in immunologic responder rates.

- Tables with similar format to Table 127:
- Table 128: ALS Responses to S. flexneri 2a LPS, Immunologic Responder Rates by Study Day and Study Group Immunology Population
- Table 129: ALS Responses to S. flexneri 2a IpaB, Immunologic Responder Rates by Study Day and Study Group Immunology Population
- Table 130: ALS Responses to S. flexneri 2a IpaC, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 131: ALS Responses to S. flexneri 2a IpaD, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 132: ALS Responses to S. sonnei Invaplex, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 133: ALS Responses to S. sonnei LPS, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 134: ALS Responses to S. sonnei IpaB, Immunologic Responder Rates by Study Day and Study Group Immunology Population
- Table 135: ALS Responses to S. sonnei IpaC, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 136: ALS Responses to S. sonnei IpaD, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

Table 137: Fecal IgA Responses to S. flexneri 2a Invaplex, Immunologic Responder Rates by Study Day and Study Group -**Immunology Population** 

| | | 4 L 22.02 | Group 1B, | Group 1B, | A C 21107 | Group 2B, | Group 2B, | |
|---|---|---|---|---|---|---|---|---|
| I ime Point | Statistic | Group 1A | Naïve | Veteran | Group 2A | Naïve | Veteran | P-Value <sup>1</sup> |
| | | $(\mathbf{v} - \mathbf{v})$ | (N=X) | (N=X) | (V-VI) | (N=X) | (N=X) | |
| Day 4 | n | XX | | | | | | |
| | Responder % | XX.X | | | | | | X.XXXX |
| | 95% CI | XX.X, XX.X | | | | | | |
| Day 8 | u | | | | | | | |
| ı | Responder % | | | | | | | |
| ı | 95% CI | | | | | | | |
| Day 15 | n | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 29 | n | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |

IgA: Immunoglobulin A; N: Number of subjects in the immunogenicity population; n: Number of subjects with data at the specified time point; Responder defined as ≥4-fold increase in titer from baseline; CI: Exact Clopper-Pearson Confidence Interval

Tables with similar format to Table 137:

Table 138: Fecal IgA Responses to S. flexneri 2a LPS, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

Table 139: Fecal IgA Responses to S. flexneri 2a IpaB, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

Table 140: Fecal IgA Responses to S. flexneri 2a IpaC, Immunologic Responder Rates by Study Day and Study Group -Immunology Population Table 141: Fecal IgA Responses to S. flexneri 2a IpaD, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

P-values are from Fisher's exact 2-tailed tests of differences between groups in immunologic responder rates.

- Table 142: Fecal IgA Responses to S. sonnei Invaplex, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 143: Fecal IgA Responses to S. sonnei LPS, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 144: Fecal IgA Responses to S. sonnei IpaB, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 145: Fecal IgA Responses to S. sonnei IpaC, Immunologic Responder Rates by Study Day and Study Group -**Immunology Population**
- Table 146: Fecal IgA Responses to S. sonnei IpaD, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

Table 147: Salivary IgA Responses to S. flexneri 2a Invaplex, Immunologic Responder Rates by Study Day and Study Group -Immunology Population

| | • | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | Group 1A<br>(N=X) | Group 1B,<br>Naïve<br>(N=X) | Group 1B, Veteran (N=X) | Group 2A<br>(N=X) | Group 2B,<br>Naïve<br>(N=X) | Group 2B, Veteran (N=X) | P-Value <sup>1</sup> |
| Day 2 | u | XX | | | | | | |
| | Responder % | XX.X | | | | | | X.XXXX |
| | 95% CI | XX.X, XX.X | | | | | | |
| Day 4 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 6 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 8 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 15 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 29 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| Day 57 | u | | | | | | | |
| | Responder % | | | | | | | |
| | 95% CI | | | | | | | |
| IgA: immunoglo | IgA: immunoglobulin A; N: number of subjects in the immunogenicity population; n: number of subjects with data at the specified time point; Responder defined | subjects in the imi | nunogenicity popu | ılation; n: number | of subjects with da | ata at the specified | time point; Respo | nder defined |

as ≥4-fold increase in titer from baseline; CI: Exact Clopper-Pearson Confidence Interval

¹P-values are from Fisher's exact 2-tailed tests of differences between groups in immunologic responder rates.

Version 1.0; 04OCT2023

# Tables with similar format to Table 147:

- Table 148: Salivary IgA Responses to S. flexneri 2a LPS, Immunologic Responder Rates by Study Day and Study Group - Immunology Population
- Table 149: Salivary IgA Responses to S. flexneri 2a IpaB, Immunologic Responder Rates by Study Day and Study
   **Group - Immunology Population**
- Table 150: Salivary IgA Responses to S. flexneri 2a IpaC, Immunologic Responder Rates by Study Day and Study **Group - Immunology Population**
- Table 151: Salivary IgA Responses to S. flexneri 2a IpaD, Immunologic Responder Rates by Study Day and Study Group - Immunology Population
- Table 152: Salivary IgA Responses to S. sonnei Invaplex, Immunologic Responder Rates by Study Day and Study **Group - Immunology Population**
- Fable 153: Salivary IgA Responses to S. sonnei LPS, Immunologic Responder Rates by Study Day and Study Group **Immunology Population**
- Table 154: Salivary IgA Responses to S. sonnei IpaB, Immunologic Responder Rates by Study Day and Study Group **Immunology Population**
- Table 155: Salivary IgA Responses to S. sonnei IpaC, Immunologic Responder Rates by Study Day and Study Group -Immunology Population
- Table 156: Salivary IgA Responses to S. sonnei IpaD, Immunologic Responder Rates by Study Day and Study Group -**Immunology Population**

### 16 References

- 1. Crane, J.K., et al., Regulation of intestinal guanylate cyclase by the heat-stable enterotoxin of Escherichia coli (STa) and protein kinase C. Infect Immun, 1992. **60**(12): p. 5004-12.
- 2. Das, J.K., et al., *Vaccines for the prevention of diarrhea due to cholera, shigella, ETEC and rotavirus.* BMC Public Health, 2013. **13 Suppl 3**: p. S11.
- 3. Pasetti, M.F., et al., *Immunology of gut mucosal vaccines*. Immunol Rev, 2011. **239**(1): p. 125-48.
- 4. Riddle, M.S., et al., *Incidence, etiology, and impact of diarrhea among long-term travelers (US military and similar populations): a systematic review.* Am J Trop Med Hyg, 2006. **74**(5): p. 891-900.
- 5. Ajene, A.N., C.L. Fischer Walker, and R.E. Black, *Enteric pathogens and reactive arthritis: a systematic review of Campylobacter, salmonella and Shigella-associated reactive arthritis.* J Health Popul Nutr, 2013. **31**(3): p. 299-307.
- 6. Connor, B.A. and M.S. Riddle, *Post-infectious sequelae of travelers' diarrhea*. J Travel Med, 2013. **20**(5): p. 303-12.
- 7. Porter, C.K., et al., *The Shigella human challenge model.* Epidemiol Infect, 2013. **141**(2): p. 223-32.
- 8. Shaughnessy, H.J., R.C. Olsson, and et al., *Experimental human bacillary dysentery;* polyvalent dysentery vaccine in its prevention. J Am Med Assoc, 1946. **132**: p. 362-8.
- 9. DuPont, H.L., et al., *The response of man to virulent Shigella flexneri 2a.* J Infect Dis, 1969. **119**(3): p. 296-9.
- 10. DuPont, H.L., et al., *Inoculum size in shigellosis and implications for expected mode of transmission*. J Infect Dis, 1989. **159**(6): p. 1126-8.
- 11. DuPont, H.L., et al., *Immunity in shigellosis. II. Protection induced by oral live vaccine or primary infection.* J Infect Dis, 1972. **125**(1): p. 12-6.
- 12. Black, R.E., et al., *Prevention of shigellosis by a Salmonella typhi-Shigella sonnei bivalent vaccine.* J Infect Dis, 1987. **155**(6): p. 1260-5.
- 13. Coster, T.S., et al., *Vaccination against shigellosis with attenuated Shigella flexneri 2a strain SC602*. Infect Immun, 1999. **67**(7): p. 3437-43.
- 14. Harro, C.e.a. Shigella flexneri 2a Invaplex 50 intranasal vaccine phase 2b challenge study. in 5th International Vaccines for Enteric Diseases Conference. 2009. Malaga, Spain.
- 15. Kotloff, K.L., et al., Evaluation of the safety, immunogenicity, and efficacy in healthy adults of four doses of live oral hybrid Escherichia coli-Shigella flexneri 2a vaccine strain EcSf2a-2. Vaccine, 1995. 13(5): p. 495-502.
- 16. Levine, M.M., et al., *Pathogenesis of Shigella dysenteriae 1 (Shiga) dysentery*. J Infect Dis, 1973. **127**(3): p. 261-70.
- 17. Samandari, T., et al., *Production of IFN-gamma and IL-10 to Shigella invasins by mononuclear cells from volunteers orally inoculated with a Shiga toxin-deleted Shigella dysenteriae type 1 strain.* J Immunol, 2000. **164**(4): p. 2221-32.
- 18. Talaat, K.e.a. Flexyn2a, a candidate bioconjugate vaccines against Shigella flexneri 2a induces protective immune response in a controlled human infection model. in Vaccines for Enteric Diseases. 2017. Albufeira, Portugal.
- 19. Kaminski, R.W., et al., *Consensus Report on Shigella Controlled Human Infection Model: Immunological Assays*. Clin Infect Dis, 2019. **69**(Suppl 8): p. S596-S601.

| n Infectior<br>595. | ntrolled Human<br>8): p. S591-S59 | n <i>Shigella C</i><br>019. <b>69</b> (Sup | us Report of | al., <i>Consens</i><br>oints. Clin I | nan, C.A., et a | MacLenna Model: Cl | 20. |
|---|---|---|---|---|---|---|---|